CLINICAL TRIAL: NCT01350778
Title: Evaluation of Effectiveness and Safety of BIOMATRIX in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: Evaluation of Effectiveness and Safety of BIOMATRIX Stent (IRIS-BIOMATRIX)
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Dio (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: CVRF2010-03
Record Dates: First submitted 2011-05-04; First posted 2011-05-10 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease requiring drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Biomatrix stent: patients treated with Biomatrix stent

SUMMARY:
The objective of this study is to evaluate effectiveness and safety of BioMatrix stent in the "real world" daily practice as compared with first-generation drug-eluting stents (sirolimus- or paclitaxel-eluting stents).

DETAILED DESCRIPTION:
This study is a non-randomized, prospective, open-label registry to compare the efficacy and safety of BioMatrix stents versus first-generation drug-eluting stent (DES) in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving BioMatrix stents
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Patients with a mixture of other DESs
* Terminal illness with life expectancy <1 year
* Patients with cardiogenic shock

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving BioMatrix stents
Sampling Method: Non-Probability Sample
Enrollment: 837 (Actual)
Dates: Start 2010-05; Primary Completion 2016-07-01 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
composite of death, nonfatal myocardial infarction (MI), or ischemic-driven Target- Vessel Revascularization (TVR) | 12 months post procedure

SECONDARY OUTCOMES:
All Death | one month
All Death | 6 months
All Death | yearly upto 5 years
Cardiac death | one month
Cardiac death | 6 months
Cardiac death | yearly upto 5 years
MI | one month
MI | 6 months
MI | yearly upto 5 years
Composite of death or MI | one month
Composite of death or MI | 6 months
Composite of death or MI | yearly upto 5 years
Composite of cardiac death or MI | one month
Composite of cardiac death or MI | 6 months
Composite of cardiac death or MI | yearly upto 5 years
TVR | one month
TVR | 6 months
TVR | yearly upto 5 years
Target-lesion revascularization (TLR) | one month
Target-lesion revascularization (TLR) | 6 months
Target-lesion revascularization (TLR) | yearly upto 5 years
Stent thrombosis (ARC criteria) | one month
Stent thrombosis (ARC criteria) | 6 months
Stent thrombosis (ARC criteria) | yearly upto 5 years
Procedural success defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization | 3 days in average
  At discharge from the index hospitalization, participants will be followed for the duration of hospital stay, an expected average of 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center; Ki Bae Seung, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital, Catholic University of Korea
Locations (20):
- South Korea (20):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - National Health Insurance Corporation Ilsan Hospital, Ilsan
  - Gachon University Gil Hospital, Incheon
  - Inha University Hospital, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Kwangju Christian Hospital, Kwangju
  - Dong-A Medical Center, Pusan
  - Inje University Pusan Paik Hospital, Pusan
  - Asan Medical Center, Seoul
  - Eulji general hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea St. Paul's Hospital, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si